CLINICAL TRIAL: NCT04406844
Title: An Observational Study to Identify the Issues and Challenges in Cancer Patients on Active Treatment During the COVID-19 Pandemic and the Resulting Lockdown
Brief Title: Issues and Challenges in Cancer Patients on Active Treatment During the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: Onco_Covid-19
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Oncology Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In view of increasing cases of SARS-CoV-2 leading to the COVID-19 Pandemic in India,there has been unprecedented restrictions on travel, work and other aspects of daily life. Our study has been designed to collect data of cancer patients to analyze their issues and challenges during Covid-19 Pandemic.

DETAILED DESCRIPTION:
Protocol No: Onco_Covid-19

Version no:1.0

Objectives: Firstly the patients recently diagnosed with cancer will be selected for enrollment who are on active treatment during lockdown based on the date of their registration in the hospital. This is followed by a telephonic interview with patients or their attendant to carry out a prospective, cross-sectional, observational study in order to address the issues and challenges faced by them during Lockdown.

Collection of data will be done through telephonic communication. Participation in this study will be entirely voluntary. Telephonic verbal consent will be taken from the patients or their attendants before collection of their response on the study questionnaire and then will be asked questions accordingly based on the questionnaire which is available in English and Hindi both. Data and general information regarding participants will only be collected in questionnaire. No personal data of the participants will be taken which will also be conveyed to the participant or attendant during telephonic verbal consent.

ELIGIBILITY:
Inclusion Criteria:

* Registered with the Max Institute of Cancer Care between Nov 1st 2019 to Jan 31st 2020
* Were scheduled to receive one or more modalities of treatment (chemotherapy, surgery, radiation therapy, immunotherapy) during the period Feb 1st 2020 to April 30th 2020

Exclusion Criteria:

-

Ages: 12 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise all the cancer patients who are registered in the Max Superspeciality hospital, Patparganj between Nov 1st 2019 to Jan 31st 2020
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-09 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Oncology patients | 4-8 weeks
  To focus on basic issues encountered by oncology patients such as transportation, medical facility, healthcare support, disease apprehension etc

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Kadayaprath, Principal Investigator — Max Hospital, Patparganj
Locations (1):
- Max Superspeciality hospital, A Unit of Balaji Medical and Diagnostic Centre, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing protocol is undecided at this stage. We may, however, provide the data if requested.